CLINICAL TRIAL: NCT00324831
Title: Phase III, Double-Blind, Randomized, Placebo-Controlled Trial of FavID® (Id/KLH) and GM-CSF Following CHOP/Rituximab as First-Line Therapy in Subjects With High-Intermediate and High-Risk Diffuse Large B-Cell Lymphoma
Brief Title: GM-CSF With or Without Vaccine Therapy After Combination Chemotherapy and Rituximab as First-Line Therapy in Treating Patients With Stage II, Stage III, or Stage IV Diffuse Large B-Cell Lymphoma
Status: Suspended | Phase: Phase 3 | Type: Interventional
Sponsor: Favrille (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000466677; FAV-ID-11; FAV-WIRB-20051774
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-03

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Doxorubicin; Prednisone; Rituximab; sargramostim; Vincristine; Methods; Immunization, Passive; Biological Therapy; Drug Therapy; Antibodies, Monoclonal; Coal Tar; Immunotherapy, Active

INTERVENTIONS:
Drug: autologous immunoglobulin idiotype-KLH conjugate vaccine
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: rituximab
Drug: sargramostim
Drug: vincristine
Procedure: Intervention/procedure
Procedure: antibody therapy
Procedure: biological therapy
Procedure: chemotherapy
Procedure: colony-stimulating factor therapy
Procedure: cytokine therapy
Procedure: monoclonal antibody therapy
Procedure: non-specific immune-modulator therapy
Procedure: therapeutic procedure
Procedure: tumor cell derivative vaccine
Procedure: vaccine therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Vaccines made from a person's cancer cells may help the body build an effective immune response to kill cancer cells. It is not yet known whether giving GM-CSF together with vaccine therapy is more effective than giving GM-CSF together with a placebo when given after combination chemotherapy and rituximab in treating diffuse large B-cell lymphoma.

PURPOSE: This randomized phase III trial is studying GM-CSF and vaccine therapy to see how well they work compared to GM-CSF and placebo when given after combination chemotherapy and rituximab as first-line therapy in treating patients with stage II, stage III, or stage IV diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the 3-year disease-free survival of patients with high-intermediate- or high-risk bulky stage II or stage III or IV diffuse large B-cell lymphoma treated with sargramostim (GM-CSF) with or without autologous immunoglobulin idiotype-KLH conjugate vaccine (FavId®) after combination chemotherapy comprising cyclophosphamide, doxorubicin, vincristine, prednisone, and rituximab (CHOP-R).

Secondary

* Compare the 2-year disease-free survival, duration of response, time to progression, overall survival, and safety in patients treated with these regimens.
* Estimate the rate of immune reactivity to FavId®.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to risk score (3 [high-intermediate] vs 4 or 5 [high]).

* Chemotherapy: Patients receive cyclophosphamide IV, doxorubicin hydrochloride IV, vincristine IV, and rituximab IV on day 1 and oral prednisone on days 1-5. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
* Sargramostim (GM-CSF) with or without autologous immunoglobulin idiotype-KLH conjugate vaccine (FavId®): Patients achieving complete remission (CR) or unconfirmed CR after chemotherapy and who have FavId® available are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive FavId® vaccine subcutaneously (SC) on day 1. Patients also receive sargramostim (GM-CSF) SC on days 1-4.
  * Arm II: Patients receive placebo SC on day 1 and GM-CSF SC as in arm I. In both arms, treatment repeats once a month for 6 months and then once every 2 months for 24 months (18 total vaccinations) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 2 years.

PROJECTED ACCRUAL: A total of 480 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diffuse large B-cell lymphoma

  * Bulky stage II or stage III or IV disease
  * Treatment naïve
  * International Prognostic Index score of 3 (high-intermediate) or 4/5 (high)
* Lymphoma accessible for sampling or existing biopsy material judged suitable for preparation of autologous immunoglobulin idiotype-KLH conjugate vaccine (FavId®)
* No history of CNS lymphoma or meningeal lymphomatosis
* No history of indolent lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Platelet count > 75,000/mm^3
* ALT and AST < 2 times upper limit of normal
* Not pregnant or nursing
* No history of unresolved hepatitis B viral infection
* No history of a treated prior malignancy unless in remission ≥ 2 years, except for treated nonmelanoma carcinomas of the skin or in situ cervical carcinomas or prostatic carcinomas
* No contraindication to doxorubicin hydrochloride (e.g., abnormal contractility on ECG)
* No contraindication to vincristine (e.g., peripheral neuropathy)
* No know HIV positivity
* No serious nonmalignant disease, including any of the following:

  * Psychiatric disorders
  * Compromised pulmonary function
  * Congestive heart failure
  * Active bacterial, viral, or fungal infections

PRIOR CONCURRENT THERAPY:

* No prior keyhole limpet hemocyanin
* No planned radiotherapy during or after study therapy
* No concurrent systemic immunosuppressive therapy (e.g., steroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival as measured by the Kaplan-Meier method at 3 years

SECONDARY OUTCOMES:
Disease-free survival as measured by the Kaplan-Meier method at 2 years
Duration of response (complete or partial response)
Overall disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: John F. Bender, PharmD, Study Chair — Favrille
Locations (2):
- United States (2):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina